CLINICAL TRIAL: NCT06856096
Title: PET/MRI Artificial Intelligence Reconstruction Algorithm AIR Recon DL Image Quality Evaluation and Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20252044
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Parkinson's Syndrome
Keywords: Artificial Intelligence Reconstruction Algorithms; AIR Recon DL; PET/MRI

STUDY DESIGN:
Intervention Model Description: Comparison between different patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Comparison between different patients (Experimental): This is a diagnostic pilot study in which 50 patients with disorders of consciousness, Parkinson's syndrome and 15 prostate cancer patients were recruited to undergo PET/MRI imaging to evaluate the impact of AIR Recon DL on scanning and imaging time in different diseases and imaging sites, to determine its efficiency in clinical applications and to analyse its potential advantages in the diagnosis of specific diseases.
  Interventions: Diagnostic Test: PET/MRI

INTERVENTIONS:
Diagnostic Test: PET/MRI — PET/MR imaging using an integrated TOF PET/MR scanner (Signa, GE Healthcare, WI, USA)

SUMMARY:
PET/MRI artificial intelligence reconstruction algorithm AIR Recon DL image quality evaluation and clinical study

DETAILED DESCRIPTION:
This is a diagnostic pilot study in which 50 patients with disorders of consciousness, Parkinson's syndrome and 15 prostate cancer patients were recruited to undergo PET/MRI imaging to evaluate the impact of AIR Recon DL on scanning and imaging time in different diseases and imaging sites, to determine its efficiency in clinical applications and to analyse its potential advantages in the diagnosis of specific diseases.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults between the ages of 18 and 75 who are autonomous; 2. persons with good compliance; 3. those who are mentally alert and able to move around on their own; 4. Those who agree to participate in this clinical trial and sign the informed consent form.

Exclusion Criteria:

* 1. Persons who do not have full capacity for civil behaviour; 2. Women during pregnancy and breastfeeding; 3. other implants, prostheses, foreign bodies and patches with electronic implants such as pacemakers, insulin pumps and cochlear implants that are not suitable for MRI; 4. patients with claustrophobia; 5. those who, in the opinion of the investigator, are not suitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Signal to Noise Ratio | 1 day from injection of the tracer
  An important parameter for measuring image quality, indicating the ratio of signal to noise power
Contrast to Noise Ratio | 1 day from injection of the tracer
  Describes the relative difference in signal strength between the two tissues, the greater the difference the better the image comparison

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine,Xijing Hospital, Fourth Military Medical University, Xi'an, China, Xi'an, Shaanxi Province, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No